CLINICAL TRIAL: NCT05470452
Title: Validating the Safety and Effectiveness of ENDOANGEL Upper Gastrointestinal Endoscope Image Auxiliary Diagnostic Software
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: The Second Affiliated Hospital of Chongqing Medical University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Diagnostic
Other Study IDs: EndoAngel -CTP-02
Record Dates: First submitted 2022-07-20; First posted 2022-07-22 (Actual); Last update posted 2022-07-22 (Actual); Status verified 2022-07

CONDITIONS: Gastric Cancer
MeSH Terms: conditions — Stomach Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Physician AI-assisted diagnosis group (Experimental)
  Interventions: Other: The reading process is assisted by ENDOANGEL
- Physician Independent Diagnostic Group (Sham Comparator)
  Interventions: Other: No ENDOANGEL assistance during the reading process

INTERVENTIONS:
Other: The reading process is assisted by ENDOANGEL — Diagnosis of benign and malignant lesions with the help of ENDOANGEL
  Arms: Physician AI-assisted diagnosis group
Other: No ENDOANGEL assistance during the reading process — Diagnosis of benign and malignant lesions without the help of ENDOANGEL
  Arms: Physician Independent Diagnostic Group

SUMMARY:
The upper Gastrointestinal Endoscope Image Auxiliary Diagnostic Software developed by Wuhan ENDOANGEL Medical Technology Co., Ltd. is used for the identification of gastric cancer in endoscopic magnification mode in definitive images to assist in the diagnosis of upper gastrointestinal gastric cancer lesions. The aim of this study is to evaluate the safety and effectiveness of the software in clinical use.

ELIGIBILITY:
Inclusion Criteria:

1. Age ≥18, male or female；
2. Cases with complete, clear imaging data, including images under white light and magnified stained images；
3. Complete pathological diagnosis of upper digestive tract lesions;
4. The included cases were excluded from the software development.

Exclusion Criteria:

1. Cases whose image data did not meet the evaluation requirements;
2. The investigator considered the case unsuitable for the clinical trial.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 340 (Estimated)
Dates: Start 2021-07-28 (Actual); Primary Completion 2022-08 (Estimated); Study Completion 2022-08 (Estimated)

PRIMARY OUTCOMES:
AFROC-AUC | 3 months
  AFROC-AUC at the level of identified lesions in the upper gastrointestinal cancers in the trial and control groups, using a between-group comparison.

SECONDARY OUTCOMES:
Cancer identification Sensitivity | 3 months
  The numerator is the number of true positives and the denominator is the total number of true positives and false negatives.
Cancer identification specificity | 3 months
  The numerator is the number of true negatives and the denominator is the total number of true negatives and false positives.
Cancer Identification Diagnosis Compliance Rate | 3 months
  The numerator is the total number of true positives plus true negatives, and the denominator is the total number of true positives, false positives, true negatives, and false negatives.

CONTACTS AND LOCATIONS:
Locations (1):
- The Second Hospital of Chongqing Medical University, Chongqing, Chongqing Municipality, China